CLINICAL TRIAL: NCT05543590
Title: Effect of Plasmapheresis on Clinical Improvement and Biological Parameters of Patients With Long-haul COVID: PLEXCOVIL Study, a Randomized Controlled Study.
Brief Title: Effect of Plasmapheresis on Clinical Improvement and Biological Parameters of Patients With Long-haul COVID
Acronym: PLEXCOVIL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-
Record Dates: First submitted 2022-07-26; First posted 2022-09-16 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Long-Haul COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Plasmapheresis; Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: receiving plasmapheresis (Experimental)
  Interventions: Drug: Plasmapheresis; Other: Blood collection; Other: Stool samples; Other: PET scan; Other: Cycle ergometer stress test; Other: Questionnaires at baseline
- Control group : no treatment (Other)
  Interventions: Other: Blood collection; Other: Stool samples; Other: PET scan; Other: Cycle ergometer stress test; Other: Questionnaires at baseline; Other: Medical consultations

INTERVENTIONS:
Drug: Plasmapheresis — 5 sessions of plasma exchanges
  Arms: Experimental group: receiving plasmapheresis
Other: Blood collection — Blood collection to assess biological markers at baseline, M3 and M12
Other: Stool samples — Stool samples will be collected from participants at baseline,M3 and M12
Other: PET scan — PET scan at baseline and M6
Other: Cycle ergometer stress test — Cycle ergometer stress test at M6
Other: Questionnaires at baseline — Questionnaires at baseline, M3 and M6
Other: Medical consultations — Medical consultations
  Arms: Control group : no treatment

SUMMARY:
Many patients infected with SARS-Cov-2 present in the months following infection with non-specific symptoms such as non-resolving fatigue, cognitive disorders, dyspnea, headaches, myalgias, sleep disorders, anosmia/ ageusia and post exertion malaise. The persistence of these symptoms is called "post covid syndrome" or "long Covid".

According to the literature, the pathophysiological mechanisms involved in post-covid syndromes would include an inadequate immune response, activation of autoimmunity, persistence of pro-inflammatory biomarkers, endothelial dysfunction and alterations in the intestinal microbiota.

In view of the involved pathophysiological mechanisms, linked to the circulation of pro-inflammatory molecules, autoimmunity or endothelial activation, the role of immuno-modulation in the treatment of long Covid need to be evaluated.

Plasma exchange (PE) by decreasing blood levels of pro-inflammatory cytokines and/or autoimmune markers results in moderate to marked clinical improvement in various types of autoantibody-associated inflammatory, autoimmune and neurological diseases.

The goal of our study is to evaluate the effects of plasmapheresis in patients with moderate to severe long-term COVID compared to patients receiving no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Who have had confirmed SARS-COV2 infection (RT PCR) for at least 6 months
* Having for more than 6 months at least 3 symptoms among the following: fatigue, post effort malaise, dyspnea, headache, diffuse myalgia/arthromyalgia, neuropathic pain, cognitive disorders, anosmia/ageusia
* Whose above symptoms have an impact on daily activities
* And/or on sick leave for more than 3 months
* And/or having to take to bed for more than 2 hours a day
* Having given free and informed written consent
* Being affiliated with or benefiting from social security

Exclusion Criteria:

* With suspected Covid-19 but not confirmed by RT-PCR test
* Having a known history of any other pathology that could be confused with the diagnosis of long COVID: multiple sclerosis, autoimmune disease (lupus and Gougerot syndrome, inflammatory muscle disease, and myasthenia gravis), untreated hypothyroidism, major depression, use of narcotics regular.
* Unable to perform a cycle ergometer stress test
* With innate or drug-induced coagulation disorders (oral or parenteral anticoagulation)
* With contraindications to plasmapheresis such as: lack of peripheral venous access or unstable cardiac pathology
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose fatigue has decreased by 30% on the Chalder scale at M3 compared to its initial state measured at baseline | 3 months

SECONDARY OUTCOMES:
Observation of the evolution of the fatigue (Chalder scale) felt by the patients during the 6 months of the study in the two groups of patients | 6 months
Evaluation of the quality of life (SF-36) of patients at month 3 and month 6 | 3 months and 6 months
Evaluation of the overall impression of change of patients at month 3 and month 6 (PGIC scale) | 3 months and 6 months
Evolution at month 3 and month 6 of the following clinical signs: post-exertional malaise, dyspnea, headache, myalgia, neuropathic pain, cognitive impairment, anosmia/ageusia, anxiety/depression | 3 months and 6 months
Assessment of patients' functional status at month 3 and month 6 (Post-COVID-19 functional status scale) | 3 months 6 months
Evaluation of the professional or student activity at month 3 and month 6 | 3 months and 6 months
Percentage of patients with 25% improvement in neuromuscular activity of M wave abnormalities at month 6 compared to baseline | 6 months
Percentage of patients with improved brain and/or spinal cord metabolism at month 6 compared to baseline | 6 months
Evolution of cytokine profiles and lymphocyte activation markers at month 3 and month 6 | 3 months and 6 months
Rate and evolution of autoimmune markers at month 3 and month 6 | 3 months and 6 months
Level and evolution of endothelial activity markers at month 3 and month 6 | 3 months and 6 months
Evaluation of the microbiotic signature at month 3 and month 6 | 3 months and 6 months

IPD SHARING:
Plan to Share IPD: No